CLINICAL TRIAL: NCT06746740
Title: Developing and Testing a Trauma-Informed Exercise Intervention for Women Veterans With Histories of Sexual Violence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5308-W; is 1IK2RX005308-01A1 (Other Grant/Funding Number: VA Rehabilitation Research and Development)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Sexual Violence
Keywords: women Veterans; sexual violence; exercise; transdiagnostic
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Pilot open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise (Experimental): Exercise intervention
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Adapted with input from phase 1

SUMMARY:
Exposure to sexual violence disproportionally impacts women Veterans and can have profound negative impacts on daily functioning. Current treatments for sexual violence focus on psychiatric symptoms and ignore frequently co-occurring physical and psychosocial concerns. Exercise can improve trauma-related physical, mental, and psychosocial health conditions and may help women who have experienced sexual violence. Yet, women Veterans experience many barriers to participating in exercise and prefer interventions that are tailored to their preferences. This proposal will develop and test an exercise intervention tailored specifically to women Veterans who have experienced sexual violence. Treatment development will be informed by women Veterans with histories of sexual violence and their providers. Feasibility and acceptability will be tested, and outcomes will be explored to inform future research. This intervention is urgently needed to address gaps in integrative care and persistent trauma-related health concerns among women Veterans with histories of sexual violence.

DETAILED DESCRIPTION:
Women Veterans (WVs) disproportionately experience sexual violence (SV) throughout their lifetime. These experiences of SV are often repeated, resulting in a lifelong pattern of SV victimization which can have profound negative impacts on physical, mental, and psychosocial functioning and quality of life. Current VHA policies highlight the need for integrative interventions which effectively address the diverse negative health sequelae associated with lifetime SV. Yet, there is currently a gap in treatment offerings that address broad psychiatric, physical, and psychosocial health impacts of SV. Exercise has been shown to improve trauma-related mental health conditions among survivors of SV and improve trauma-related multimorbidity among Veterans with a PTSD diagnosis. Yet, many barriers exist to exercise among WVs which contribute to low exercise engagement from this group. This Career Development Award (CDA-2) thus aims to develop and test a trauma-informed telehealth exercise intervention tailored for WVs with histories of SV. Treatment development will be guided by 1) previous interventions completed among Veterans with PTSD, 2) documented preferences among women with histories of SV, and 3) trauma-informed approaches and integration of stakeholder feedback. During phase one of this project, the investigators will conduct pre-implementation stakeholder interviews with WVs with histories of SV and related healthcare providers to provide guidance on the structure and content of the proposed intervention. This information will be used to create the program manual for the proposed intervention. During phase two of this project, WVs aged 21-65 with lifetime history of SV will be recruited to participate in an open trial consisting of a 12-week, online physical activity program including aerobic and strength training. Qualitative data will be collected in parallel with quantitative outcomes to assesses the primary feasibility and acceptability outcomes. Exploratory outcomes will include functional status. Candidate outcomes to be assessed include physical, mental, and psychosocial health outcomes. This pilot trail will extend the understanding for trauma-informed exercise approaches for WVs with histories of SV and of the feasibility, acceptability, and potential benefits of exercise for this group. Results will be used to develop a fully powered randomized controlled trial for WVs with histories of SV.

ELIGIBILITY:
Inclusion Criteria:

* Veteran self-identifies as woman
* has a history of sexual violence at any point in their lifetime
* between the ages of 21 an 65
* currently does not meet physical activity level guidelines
* reports some functional difficulties that indicate some interference in daily life
* safe and private location to engage in the virtual exercise program

Exclusion Criteria:

* does not identify a safe and private location for exercise participation
* severe drug or alcohol use disorder within the past year
* clinically significant:

  * neurological disorder
  * systemic illness affecting central nervous system function
  * history of seizure disorder in the past 5 years
  * uncontrolled diabetes
  * end stage liver disease or currently receiving dialysis
  * physical disabilities precluding use of exercise equipment
  * significant cognitive impairment
  * active signs and symptoms of CVD
  * metabolic
  * renal disease
  * if taking antidepressants must have stable regimen
  * if in psychotherapy maintain therapy throughout trial

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self-identifies as woman
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - recruitment interest | through study completion, an average of one year
  ratio interested of those approached for the workshop
feasibility, enrollment rate | through study completion, an average of one year
  Ratio enrolled (consented) of those approached
feasibility qualitative via Narrative Evaluation of Intervention Interview | Through study completion, an average of 3 months.
  Identification of challenges and facilitators during the recruitment process as assessed by study staff as well as feedback from focus group participants generated using the Narrative Evaluation of Intervention Interview (NEII). This is an interview composed of 16 open ended questions that allows participants to evaluate the process and outcomes of the intervention. Reviewers will generate a list of themes based on the responses to this interview.
acceptability - Veteran adherence | Through study completion, an average of one year.
  Attendance rate for the 12-week intervention
Acceptability- Quantitative satisfaction via Client satisfaction questionnaire Change | assessed at BL, 12 weeks, 24 week follow up
  Client satisfaction questionnaire (CSQ-8), total scores range from 8 to 32 with higher scores indicating higher satisfaction.

SECONDARY OUTCOMES:
Functional Status - The World Health Organization Disability Assessment Schedule 2.0 (WHODAS-2) | baseline, post-intervention (12 weeks), follow up (24 weeks)
  The World Health Organization Disability Assessment Schedule 2.0 (WHODAS-2) is a 36-item self-report tool that assesses functioning in the past 30 days among six specific domains (i.e., cognition, physical mobility, self-care, social, domestic/occupational, and participation in society) and provides an overall disability score. Higher scores indicate greater disability
Physical Function - arm curls | baseline, post-intervention (12 weeks), follow up (24 weeks)
  number of curls in 30 seconds
Physical Activity Level - Godin Leisure-Time Exercise Questionnaire (GLTEQ) | baseline, post-intervention (12 weeks), follow up (24 weeks)
  The Godin Leisure-Time Exercise Questionnaire (GLTEQ) is a validated brief inventory assessing activity domains and aerobic activity in a typical week. Duration in minutes of exercise multiplied by number of times per week, in the past 7 days. Total minutes per week calculated; mean reported.
PTSD - PTSD Checklist-5 (PCL-5) for DSM-V | baseline, post-intervention (12 weeks), follow up (24 weeks)
  The PTSD Checklist-5 (PCL-5) for DSM-V is a 20-item self-report measure that assesses the extent to which an individual is bothered by each PTSD symptom during the past month using a 5-point Likert-type scale. Higher scores indicating more severe symptoms
Anxiety - Depression Anxiety and Stress Scale (DASS 21) | baseline, post-intervention (12 weeks), follow up (24 weeks)
  Depression Anxiety and Stress Scale (DASS 21) provides scores for depression, anxiety, and stress subscales, with higher scores indicating worse outcomes. Each item is scored on a 4-point scale (0 = Did not apply to me at all, to 3 = Applied to me very much or most of the time)
Depression - Patient Health Questionnaire (PHQ-9) | baseline, post-intervention (12 weeks), follow up (24 weeks)
  Will be assessed with the 9-item Patient Health Questionnaire. The total score can range from 0 to 27. Higher scores indicate greater severity of depression.
Psychosocial function- The Brief Inventory of Psychosocial Functioning (IPF-Brief) | baseline, post-intervention (12 weeks), follow up (24 weeks)
  Participants rank each of the 7 statements based on their overall experience over the past month on a scale from 0 (not at all) to 6 (very much). 7 is marked if the statement is not applicable. Higher scores indicate more impaired psychosocial functioning.
Pain - Short-Form McGill Pain Questionnaire | baseline, post-intervention (12 weeks), follow up (24 weeks)
  Short-Form McGill Pain Questionnaire is an 22-item measure assess pain quality/intensity. Total score ranges from 0-45. Higher scores indicate more severe pain.
Fatigue - Multidimensional Fatigue Inventory (MFI) | baseline, post-intervention (12 weeks), follow up (24 weeks)
  is a 20-item instrument that measures dimensions of fatigue. scores range from 20 to 100 with higher scores indicating greater fatigue
Health Status - 12-Item Short Form Health Survey (SF-12) | baseline, post-intervention (12 weeks), follow up (24 weeks)
  The 12-Item Short Form Health Survey (SF-12) will be used to assess overall health. Score ranging from 0 to 100. A higher score indicating a better quality of life.
Quality of Life - The Quality of Life Scale (QOLS) | baseline, post-intervention (12 weeks), follow up (24 weeks)
  Participants answer each question on a 7 point scale. It is scored by adding up the score on each item to get a minimum potential score of 16 and a maximum total score of 112. Higher scores indicate a higher quality of life.
Exercise Motivation - Behavioral Regulation in Exercise Questionnaire (BREQ-3) | baseline, post-intervention (12 weeks), follow up (24 weeks)
  Behavioral Regulation in Exercise Questionnaire (BREQ-3) uses 23 items to measure exercise motivation types, Using a 5 point Likert scale, the maximum score is 5 which indicates a high level of that particular sub-scale of motivation, e.g. intrinsic motivation or amotivation.
Physical function - chair stands | baseline, post-intervention (12 weeks), follow up (24 weeks)
  number of chair stands in 30 seconds
physical function - balance | baseline, post-intervention (12 weeks), follow up (24 weeks)
  time balancing on one foot
physical function - 2 minute step test | baseline, post-intervention (12 weeks), follow up (24 weeks)
  number of knee raised in 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Pebole, PhD MA, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No additional IPD will be shared besides the deidentified/anonymized data set and data dictionary will be shared.